CLINICAL TRIAL: NCT02727166
Title: Efecto de Fructanos Paralelamente Hidrolizados Provenientes de Achicoria Sobre Las Sensaciones Abdominales
Brief Title: Effect of Chicory-derived Inulin on Abdominal Sensations and Bowel Motor Function
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Universitari Vall d'Hebron Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PR(AG)168/2010
Record Dates: First submitted 2016-03-18; First posted 2016-04-04 (Estimated); Last update posted 2016-04-04 (Estimated); Status verified 2016-03

CONDITIONS: Functional Gastrointestinal Disorders
Keywords: intestinal gas; functional gut symptoms; intestinal sensitivity; intestinal motility
MeSH Terms: conditions — Gastrointestinal Diseases | interventions — Inulin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Inulin 8 g/d (Experimental): Mixture of oligo- and polysaccharides composed of fructose units connected by β (2→1) links with a total number of fructose and glucose units ranging between 2 and 70.
  Interventions: Dietary Supplement: Inulin
- maltodextrine 8 g/d (Placebo Comparator)
  Interventions: Dietary Supplement: Maltodextrine

INTERVENTIONS:
Dietary Supplement: Inulin — Administered in 4 g sacchets taken in 200 mL liquid during breakfast and dinner for 4 week intervention period
  Arms: Inulin 8 g/d
Dietary Supplement: Maltodextrine — Administered in 4 g sacchets taken in 200 mL liquid during breakfast and dinner for 4 week intervention period
  Arms: maltodextrine 8 g/d

SUMMARY:
Subjects with gas-related complaints exhibit impaired handling of intestinal gas loads and we hypothesized that inulin would have a beneficial effect. Aim: to determine the effect of a prebiotic chicory-derived inulin-type fructan on the tolerance of intestinal gas. Methods. Placebo-controlled, parallel, randomized and double-blind trial study. Subjects with abdominal symptoms and reduced tolerance of intestinal gas (selected by a pre-test) will receive either inulin (8 g/d, n=18) or maltodextrin as a placebo (8 g/d, n=18) for 4 wk. A gas challenge test (4 h jejunal gas infusion at 12 mL/min while measuring abdominal symptoms and gas retention for 3 h) will be performed before and at the end of the intervention phase. Gastrointestinal symptoms and bowel habits (using daily questionnaires for 1 wk) and fecal bifidobacteria counts will be measured before and at the end of the intervention.

ELIGIBILITY:
Inclusion Criteria:

* negative sensation of digestive well-being (score ≤ 1 on at least 2 of the 6 evaluation days, scored on a - 5 / +5 scale.
* poor tolerance of a gas challenge test (abdominal perception score ≥ 3, on a 0-6 scale, for at least three 15-min time points over the last 90 minutes of the 180-minute-long intestinal gas infusion test).

Exclusion Criteria:

* antibiotic intake,
* exceptional diets,
* changes in dietary habits or intake of Ca supplements over the preceding month.

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2010-11; Primary Completion 2015-07 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Perception of intestinal gas infusion | 60 last min of the 180 min gas infusion test
  Effect of inulin intake (change from baseline with inulin versus placebo) on the tolerance of the gas challenge test, measured as the perception score of digestive sensations during the gas challenge test. At each time point, the highest score instead of the mean or cumulative scores will be computed for comparisons; these scores will be averaged over the last 60 min of the test in each subject; the differences between basal and intervention periods (inulin or placebo) will be calculated.

SECONDARY OUTCOMES:
Intestinal gas retention | 60 last min of the 180 min gas infusion test
  Effect of inulin intake (change from baseline with inulin versus placebo) on the volume of gas retention (volume infused minus volume evacuated) measured as the average value over the last 60 min of the gas infusion test.
Digestive well-being | 6 last days of intervention
  Effect of inulin intake (change from baseline with inulin versus placebo) on digestive well-being measured by daily questionnaires on - 5 to + 5 score scales and averaged over 6 days.
Abdominal discomfort | 6 last days of intervention
  Effect of inulin intake (change from baseline with inulin versus placebo) on abdominal discomfort measured by daily questionnaires on 0 to 10 score scales and averaged over 6 days.
Bowel habit | 6 last days of intervention
  Effect of inulin intake (change from baseline with inulin versus placebo) on the number of bowel movements measured by daily questionnaires during 6 days.

CONTACTS AND LOCATIONS:
Overall Officials: Fernando Azpiroz, MD, Principal Investigator — Vall d'Hebron Research Institute

IPD SHARING:
Plan to Share IPD: Undecided